CLINICAL TRIAL: NCT01400256
Title: The Use of Valsartan for the Management of Blood Pressure in Acute Stroke: Affects on Cerebral Blood Flow
Brief Title: Blood Pressure Lowering in Acute Stroke Trial
Acronym: BLAST
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment/patient population
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Neil Schwartz, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A US71
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Stroke, Acute
Keywords: diagnostic
MeSH Terms: conditions — Stroke; Disease | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Valsartan — After the initial MRI, patients will be given a 160 mg dose of valsartan or placebo, in a double-blinded fashion. A sustained MAP reduction of 15-20% will be the goal. If the MAP remains within 15% of the initial value (prior to the first MRI scan) 24 hours after the first dose of valsartan (or placebo), the patients will be given a 320 mg dose of valsartan (or placebo) and will remain on valsartan 320 mg (or placebo) daily until day 7, or hospital discharge (whichever is sooner). If the MAP is falls by more than 20% after the 160 mg (or placebo) dose, the patient will be switched to 80 mg of valsartan (or placebo) until day 7, or hospital discharge (whichever is sooner). If the blood pressure is lowered by 15-20% (the goal), the patients will remain on valsartan 160 mg (or placebo) daily for the duration of the study.

SUMMARY:
The investigators hope to show that valsartan can be used safely in the setting of acute stroke to lower elevated blood pressure. There are novel properties of this class of drug (an angiotensive-receptor blocker or ARB), and promising human and animal data, that would suggest this drug can be safely used to lower blood pressure in the setting of acute stroke without compromising brain blood flow (i.e. cerebral perfusion). If this is proved to be the case, this compound could potentially be used routinely in this setting, with the hope of improving outcome. This pilot study may pave the way for a larger randomized trial looking at outcome measures in stroke patients. Further, a positive result in the this pilot study will serve as proof of concept that ARBs maintain cerebral perfusion while decreasing blood pressure, an overall favorable property.

DETAILED DESCRIPTION:
Patients who are suffering from a stroke often present to the hospital with elevated blood pressure. Elevated blood pressure in the setting of stroke increases the risk of brain swelling or bleeding into the brain. Even so, there has been concern about lowering the blood pressure with medications because the newly injured parts of the brain may not get the blood flow they need, thereby worsening the damage from the initial stroke. We hope to demonstrate that the drug valsartan can be used to safely and modestly lower blood pressure in acute stroke patients, without having a detrimental effect on brain blood flow or neurologic status. Novel MRI techniques to measure brain blood flow will be used in conjunction with clinical scales to demonstrate safety.

We intend to enroll 20 patients (10 for active drug, 10 for placebo) over an 16 month period. Patients admitted with the diagnosis of acute stroke and hypertension will be eligible for the study. All patients will be screened by the attending physician on the Stroke Service. Informed consent will be obtained from the patient or a suitable surrogate. Baseline characteristics will be recorded including demographics, drug allergies, date and time of presumed stroke, prior stroke history, history of hypertension, current blood pressure regimen, other cardiovascular risk factors, baseline physical exam, National Institute of Health Stroke Scale (NIHSS) score, and baseline modified Rankin score. Patients will be treated and examined daily by neurologists from the Stroke Service and/or Neurocritical Care teams.

A sustained mean arterial pressure (MAP) of 110 (~150/90) or greater is needed for inclusion in the study. Upon admission, as per our usual protocol, antihypertensive medications will be withheld. In general, we do not administer antihypertensive agents to acute ischemic stroke patients unless the blood pressure is greater than ~200/110 (MAP 140) or the patient has signs or symptoms thought to be secondary to elevated blood pressure. Blood pressure will be taken at least every four hours, as per protocol, either manually or with an automated device. Mean arterial pressure (MAP) will be calculated using a standard formula (MAP = diastolic blood pressure + 1/3 pulse pressure). Patients admitted to the ICU may have arterial lines placed for continuous blood pressure monitoring, if needed as part of their routine care. Routine blood chemistries, including serum creatinine and liver function tests will be drawn prior to administering drug or placebo.

At enrollment, the patient will be randomized to receive either valsartan or placebo. The first dose of study medication will not be administered until after the baseline MRI.

The patient will undergo an initial MRI that includes diffusion-weighted imaging (DWI) and perfusion-weighted imaging (PWI). The initial MRI is standard care for stroke patients. After the initial MRI, patients will be given a 160 mg dose of valsartan or placebo, in a double-blinded fashion. A sustained MAP reduction of 15-20% will be the goal. If the MAP remains within 15% of the initial value (prior to the first MRI scan) 24 hours after the first dose of valsartan (or placebo), the patients will be given a 320 mg dose of valsartan (or placebo) and will remain on valsartan 320 mg (or placebo) daily until day 7, or hospital discharge (whichever is sooner). If the MAP is falls by more than 20% after the 160 mg (or placebo) dose, the patient will be switched to 80 mg of valsartan (or placebo) until day 7, or hospital discharge (whichever is sooner). If the blood pressure is lowered by 15-20% (the goal), the patients will remain on valsartan 160 mg (or placebo) daily for the duration of the study.

A follow-up MRI with PWI and DWI will be obtained between 48-96 hours of the initial scan. Additional antihypertensive agents will not be administered until after the follow-up MRI scan unless deemed medically indicated by the attending physician. If additional agents are administered, any antihypertensive can be used except for an ACE inhibitor or ARB. Any additional agents needed for blood pressure control will be recorded.

The patient will continue taking valsartan vs. placebo throughout the duration of his/her hospitalization. At the time of discharge, an NIHSS and modified Rankin score will be recorded. On hospital day 7, or discharge (whichever is sooner), study medication will be discontinued and blood pressure medication will be at the discretion of the treating physician.

A 30-day follow-up will include assessment of a modified Rankin score and Glasgow Outcome Score. This 30 day follow-up will be conducted by telephone unless the patient is coming to the clinic for a routine hospital follow-up visit.

The patients will undergo two brain MRIs during the initial hospitalization, each requiring a scanning time of approximately 45 minutes. Standard sequences will be obtained, including DWI and PWI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women over age 18 who have had an acute ischemic stroke referable to the anterior circulation, as diagnosed by one of more of the following: clinical judgment, head CT, and/or MR imaging [i.e. a positive diffusion-weighted imaging (DWI) abnormality].
2. Clinical syndrome not likely to represent transient ischemic attack (TIA) or other non-stroke etiology
3. Patient must be neurologically stable at the time of first MRI scan (i.e. stable NIH Stroke Scale score).
4. Initial MRI scan obtainable within 48 hours of symptom onset.
5. A pre-existing diagnosis of hypertension, either treated or untreated.
6. Average of two mean arterial blood pressures (separated by at least five minutes) at time of initial MRI scan ≥ 110.

Exclusion Criteria:

1. Patients who have taken an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) within seven (7) days of admission.
2. Patients who received intravenous or intra-arterial r-TPA for their current symptoms, or those who underwent mechanical thrombolysis.
3. Patients with hemorrhagic strokes, as seen on the initial head CT.
4. Patients with stroke-like symptoms, but no demonstrable lesion on DWI, or a DWI lesion < 2 cm in diameter (greatest dimension).
5. Patients with high-grade (>70%) internal carotid artery stenosis or occlusion ipsilateral to the current stroke.
6. Patients with high-grade aortic or mitral stenosis.
7. Patients with a previous adverse reaction to valsartan or other ARBs.
8. Patients with contraindications for MRI, including pacemakers, claustrophobia, or severe obesity.
9. Patients who are medically unstable for MR imaging, as determined by the treating team.
10. Patients with a severe co-existing disease that may interfere with the conduct of the study.
11. Patients receiving investigational drug therapies.
12. Informed consent cannot be obtained from the patient or their legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Albers, M.D, Principal Investigator — Stanford University; Neil Schwartz, M.D, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States